CLINICAL TRIAL: NCT04658875
Title: Effect of a Systematic Physical Exercise Program and Spirulina Maxima Supplementation on the Body Composition, Physical Function and Blood Lipid Profile in Sedentary Older Adults With Excess Weight
Brief Title: Effect of Spirulina Maxima and Exercise on General Fitness and Blood Lipids in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Marco Antonio Hernández Lepe, Principal Investigator, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 998/2020-2
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: evaluate the synergy presented by a supplement such as S. maxima in a systematic physical exercise program on the body composition, physical function and blood lipid profile of sedentary older adults with excess weight in a randomized, double-blind, crossover, placebo controlled trial.
  This experimental design was chosen to eliminate inter-individual differences related to Spirulina maxima/placebo
Who Masked: Participant, Investigator
Masking Description: Participants' group allocations will be performed by an independent researcher, who has not any other participation during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Spirulina maxima supplementation and exercise group (Experimental): Supplementation with Spirulina maxima (4.5 g/d) with a systematic physical exercise program during 12 weeks, then a 2 weeks washout, to finally proceed to the other treatment during 12 more weeks. During the 26 weeks of study duration every participant will have a personal isoenergetic diet.
  Interventions: Dietary Supplement: Spirulina maxima supplementation; Other: Wash-out; Other: Isoenergetic diet; Other: Systematic physical exercise program
- Spirulina maxima supplementation (Experimental): Supplementation with Spirulina maxima (4.5 g/d) without exercise program during 12 weeks, then a 2 weeks washout, to finally proceed to the other treatment during 12 more weeks. During the 26 weeks of study duration every participant will have a personal isoenergetic diet.
  Interventions: Dietary Supplement: Spirulina maxima supplementation; Other: Wash-out; Other: Isoenergetic diet
- Exercise group (Experimental): Systematic physical exercise program during 12 weeks, then a 2 weeks washout, to finally proceed to the other treatment during 12 more weeks. During the 26 weeks of study duration every participant will have a personal isoenergetic diet.
  Interventions: Other: Wash-out; Other: Placebo supplementation; Other: Isoenergetic diet; Other: Systematic physical exercise program
- Control group (Active Comparator): No systematic physical exercise program and No supplementation during 12 weeks, then a 2 weeks washout, to finally proceed to the other treatment during 12 more weeks. During the 26 weeks of study duration every participant will have a personal isoenergetic diet.
  Interventions: Other: Wash-out; Other: Placebo supplementation; Other: Isoenergetic diet

INTERVENTIONS:
Dietary Supplement: Spirulina maxima supplementation — Supplementation with Spirulina maxima (4.5 g/d) in capsules during 12 weeks.
  Arms: Spirulina maxima supplementation; Spirulina maxima supplementation and exercise group
Other: Wash-out — 2 weeks washout period to each study subject to avoid any possible carryover effect.
Other: Placebo supplementation — Supplementation with placebo (4.5 g/d) in capsules during 12 weeks.
  Arms: Control group; Exercise group
Other: Isoenergetic diet — All participants will have a personal isoenergetic diet according to their height, weight, body composition and daily physical activity during 26 weeks
Other: Systematic physical exercise program — Participants in the systematic physical exercise program groups will exercise for five days a week. The physical activity program will consist of Monday to Friday chair exercises performed during 24 weeks. The approximate exercise duration will be 40 to 50 min. Each exercise session has an initial or warm-up phase (~ 10 min), a main physical conditioning phase (~ 25 min), and a cool-down or relaxation phase (~ 10 min). The physical activities to select have a metabolic equivalent tasks (METs) considered as moderate, between 3.0 and 6.0 METs. Trained personnel will assist older adults to perform the activities, including articular flexibility using elastic bands, postural and proprioception exercises with materials such as rubber balls, wood sticks, and small sandbags. These activities will be selected according to the deterioration and joint stiffness that the participants could present.
  Arms: Exercise group; Spirulina maxima supplementation and exercise group

SUMMARY:
The global older adult population has grown more than any other age group, which could be explained by the decrease of birth rate and increase of life expectancy. The healthy life expectancy of older adult in Mexico is 65.8 years, and the population's life expectancy in general is 74.4 years, this means that the population meeting that age is at increased risk of developing some disease or dependence during approximately nine years of their life. For the population over 60 years, the three most frequent health conditions reported were hypertension (40%), diabetes (24.3%), and hypercholesterolemia (20.4%). In this sense, the search for a healthy lifestyle is necessary, which includes a healthy diet that includes supplementation with nutraceuticals and the daily practice of physical activity.

Regarding nutraceutical supplementation, the cyanobacterium Spirulina maxima (S. maxima) is an important source of proteins, carotenoids, phenolic compounds and polyunsaturated fatty acids which have been tested for diverse biological activities such as lipid lowering effects, however, existing studies of effects of S. maxima on body composition, physical function and blood lipid profile in humans, mainly in older adults, have a low level of evidence and absence of adequate experimental designs, so its value as a nutraceutical cannot be assured.

The effects of performing systematic physical exercise in older adults have been shown to have positive effects on body composition and blood lipid profile, so in the present study it is proposed to evaluate the synergy presented by a supplement such as S. maxima in a systematic physical exercise program on the body composition, physical function and blood lipid profile of sedentary older adults with excess weight in a randomized, double-blind, crossover, placebo controlled trial.

DETAILED DESCRIPTION:
According to international estimations, there will be an increase in the aging population worldwide; with projections of a growth in the population older than 60 years from 900 million in 2015 to two billion in 2050. This means that the older population will move from 12% to 22% of the global population. In Mexico, in the year 2000, people aged 60 and older represented 6.8% of the total population, and an increase of 28% was expected by the year 2050; and only in Baja California State, there were 183,577 inhabitants 65 yr. old and older (Men = 46.3%, Women = 53.7%). Data from a census in Baja California's cities of Mexicali and Tijuana municipalities in 2015, showed the highest cluster of older adults above 65 yr., especially women. In Tijuana, there were 78,019 inhabitants over 65 years; with a projected population by 2020 of 101,574, and 176,134 inhabitants by 2030. The healthy life expectancy of the Mexican older adult is 65.8 years. This means that if the population's life expectancy in general is 74.4 years, the population meeting that age is at increased risk of developing some disease or dependence during approximately nine years of their life. For the population over 60 years, the three most frequent health conditions reported were hypertension (40.0%), diabetes (24.3%) and hypercholesterolemia (20.4%). These diseases affect all body systems and prevent them from carrying out daily life activities such as walking, eating, preparing or buying food, and bathing, among others. In this sense, the search for a healthy lifestyle is necessary, which includes a healthy diet that includes supplementation with nutraceuticals and the daily practice of physical activity.

Regarding supplementation with nutraceuticals, the cyanobacterium S. maxima is an important source of antioxidants, currently associated with cardiovascular protection properties. For centuries it has been cultivated and used as a nutritional supplement due to its content of amino acids and essential fatty acids, vitamin C, vitamin E, carotenoids and phycocyanins. Recently, studies on S. maxima have focused on verifying the biological activity of its components, including hypolipidemic effects. However, most studies have been conducted in animal models, with only a few studies focused on the biological effect in humans. However, most studies have been conducted in animal models, with scarce studies focused on its effects on humans. Previous researches have shown smaller adipose depots, lower blood lipid concentrations, and lower body mass gain in mice administered with a high-fat diet and S. maxima than in an high-fat diet mice control. Some studies have found a decrease in body mass, waist circumference, plasma lipid levels, inflammation, and oxidative stress in hypertensive obese patients with S. maxima supplementation (2 g for three months). However, controlled studies focused on the effect of the administration of S. maxima and a systematic exercise program in humans, have not yet been reported.

Studies on the potential effects of nutraceutical supplements are increasing in number. There have been reported the effect of 2 g/day of S. maxima supplementation on 40 hypertension subjects in a double-blind, placebo-controlled randomized trial for three months. After the intervention, they reported a significant reduction of body weight, BMI, and blood pressure in the group supplemented with S. maxima, compared with that of the placebo group. Some investigators studied the effect of Spirulina supplementation (1 g/day) during three months on the body weight, BMI, and lipid profile in patients with dyslipidemia and reported a significant decrease in total cholesterol (TC), triglycerides (TG), and cholesterol associated with low-density lipoproteins (LDL-C).

Some Spirulina compounds can reduce the macrophages infiltration into visceral fat and prevent the accumulation of liver lipids, resulting in weight reduction, specifically body fat, and there has been proved the effect of Spirulina supplementation (2 g/day) during two months on the serum lipid profile of 15 patients affected by type II diabetes mellitus, resulting in a significant reduction of TG, TC, LDL-C, and free fatty acid in blood concentrations. By means of a better-structured trial.

Many of the beneficial effects of Spirulina are attributed to its nutritional content, but its action mechanisms are poorly understood. Some authors suggest that a possible component responsible of the S. maxima hypolipidemic effect is C-phycocyanin protein, which improves the blood lipid profile. Some authors suggest that C-phycocyanin increases endogenous enzymes activity, scavenging free radicals, and downregulates cofactors in fat metabolism like adenine dinucleotide phosphate. Spirulina hypolipidemic effects can be attributed to the fact that dietary supplementation with the cyanobacteria seems to have decreased the intestinal assimilation of cholesterol, probably because Spirulina compounds bind to bile acids in the jejunum, affecting the micellar solubility of cholesterol before suppressing the cholesterol absorption. However, these studies were conducted in animal models and therefore their results cannot be extrapolated to humans, and clinical studies conducted in humans are still very scarce and appropriate clinical trials are needed to elucidate this.

Furthermore, it is known that the practice of systematic physical exercise ameliorates the risk of hypertension, diabetes and hypercholesterolemia, physical exercise of moderate intensity has the best protective effect, mainly due to physiological adaptations. Exercise has been also included as part of multicomponent interventions targeting physical function in socioeconomically vulnerable older adults in rural communities. Korean older adults (n= 187) performed a 24-week program that included group exercise, nutritional supplementation and depression management, among other components. Physical function and depression were measured before and after the intervention, with significant improvements following the intervention. Thus, appropriate exercise programs need to be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary older adults
* BMI over 25 kg/m2
* Volunteered to participate

Exclusion Criteria:

* Presenting a chronical disease
* Drinking alcohol
* Taking diet supplements
* Presenting an impediment to practicing regular physical exercise

Elimination Criteria:

* Attendance by the subject of < 80% to the physical exercise sessions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in body composition | 26 weeks
  Change in body fat percentage by using air displacement plethysmography and of bioimpedance analysis.
Changes in functional physical condition | 26 weeks
  The functional physical condition will be evaluated with the Senior Fitness Test (SFT)

SECONDARY OUTCOMES:
Lower-body strength | 26 weeks
  The lower-body strength (SFT-LBS) will be assessed by the 30 s test of getting up and sitting down from a chair.
Changes in upper-body strength | 26 weeks
  The upper-body strength (SFT-UBS) will be evaluated by the 30 s arm curl with a dumbbell (men = 8-lb, women = 5-lb).
Changes in lower-body flexibility | 26 weeks
  Lower-body flexibility (SFT-LBF) will be assessed by the chair flexion test, where participants slowly flex the hip joint, reaching as much as possible or surpassing the toes.
Changes in upper-body flexibility | 26 weeks
  Upper-body flexibility (SFT-UBF) will be assessed by the hands test behind the back. The distance between the tips of the middle fingers will be assessed independently of the alignment of the back.
Changes in agility | 26 weeks
  Agility will assessed by the 2.44 m timed-up and go test (SFT- TUG), where participants had to get up of a chair, walk as fast as possible 2.44 m and sit down again.
Changes in aerobic resistance | 26 weeks
  Aerobic resistance will be evaluated by the 2-min standing marching test (SFT-marching), where participants had to perform as many repetitions (reps) as possible

OTHER OUTCOMES:
Change in blood lipid profile | 26 weeks
  Change in plasma triacylglycerols, total cholesterol, high density lipoproteins cholesterol, and low density lipoproteins cholesterol after each treatment by using standardized enzymatic methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical and Psychology School, Tijuana, California, Mexico

IPD SHARING:
Plan to Share IPD: No
Their acceptance will be formalized by means of informed consent, which explicitly describes their confidentiality strictly enforced.

REFERENCES:
- [Background] Boardley D, Fahlman M, Topp R, Morgan AL, McNevin N. The impact of exercise training on blood lipids in older adults. Am J Geriatr Cardiol. 2007 Jan-Feb;16(1):30-5. doi: 10.1111/j.1076-7460.2007.05353.x. PMID 17215640
- [Background] Chamorro G, Salazar M, Favila L, Bourges H. [Pharmacology and toxicology of Spirulina alga]. Rev Invest Clin. 1996 Sep-Oct;48(5):389-99. Spanish. PMID 9005517
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fenster CP, Weinsier RL, Darley-Usmar VM, Patel RP. Obesity, aerobic exercise, and vascular disease: the role of oxidant stress. Obes Res. 2002 Sep;10(9):964-8. doi: 10.1038/oby.2002.131. PMID 12226146
- [Background] Fujimoto M, Tsuneyama K, Fujimoto T, Selmi C, Gershwin ME, Shimada Y. Spirulina improves non-alcoholic steatohepatitis, visceral fat macrophage aggregation, and serum leptin in a mouse model of metabolic syndrome. Dig Liver Dis. 2012 Sep;44(9):767-74. doi: 10.1016/j.dld.2012.02.002. Epub 2012 Mar 22. PMID 22444524
- [Background] Hernandez Lepe MA, Wall-Medrano A, Juarez-Oropeza MA, Ramos-Jimenez A, Hernandez-Torres RP. [SPIRULINA AND ITS HYPOLIPIDEMIC AND ANTIOXIDANT EFFECTS IN HUMANS: A SYSTEMATIC REVIEW]. Nutr Hosp. 2015 Aug 1;32(2):494-500. doi: 10.3305/nh.2015.32.2.9100. Spanish. PMID 26268076
- [Background] Hosseini SM, Khosravi-Darani K, Mozafari MR. Nutritional and medical applications of spirulina microalgae. Mini Rev Med Chem. 2013 Jun 1;13(8):1231-7. doi: 10.2174/1389557511313080009. PMID 23544470
- [Background] Iwata K, Inayama T, Kato T. Effects of Spirulina platensis on plasma lipoprotein lipase activity in fructose-induced hyperlipidemic rats. J Nutr Sci Vitaminol (Tokyo). 1990 Apr;36(2):165-71. doi: 10.3177/jnsv.36.165. PMID 2117648
- [Background] Jang IY, Jung HW, Park H, Lee CK, Yu SS, Lee YS, Lee E, Glynn RJ, Kim DH. A multicomponent frailty intervention for socioeconomically vulnerable older adults: a designed-delay study. Clin Interv Aging. 2018 Sep 19;13:1799-1814. doi: 10.2147/CIA.S177018. eCollection 2018. PMID 30275687
- [Background] Kalafati M, Jamurtas AZ, Nikolaidis MG, Paschalis V, Theodorou AA, Sakellariou GK, Koutedakis Y, Kouretas D. Ergogenic and antioxidant effects of spirulina supplementation in humans. Med Sci Sports Exerc. 2010 Jan;42(1):142-51. doi: 10.1249/MSS.0b013e3181ac7a45. PMID 20010119
- [Background] Kata FS, Athbi AM, Manwar EQ, Al-Ashoor A, Abdel-Daim MM, Aleya L. Therapeutic effect of the alkaloid extract of the cyanobacterium Spirulina platensis on the lipid profile of hypercholesterolemic male rabbits. Environ Sci Pollut Res Int. 2018 Jul;25(20):19635-19642. doi: 10.1007/s11356-018-2170-4. Epub 2018 May 7. PMID 29736642
- [Background] Lee EH, Park JE, Choi YJ, Huh KB, Kim WY. A randomized study to establish the effects of spirulina in type 2 diabetes mellitus patients. Nutr Res Pract. 2008 Winter;2(4):295-300. doi: 10.4162/nrp.2008.2.4.295. Epub 2008 Dec 31. PMID 20016733
- [Background] Manrique-Espinoza B, Salinas-Rodriguez A, Moreno-Tamayo KM, Acosta-Castillo I, Sosa-Ortiz AL, Gutierrez-Robledo LM, Tellez-Rojo MM. [Health conditions and functional status of older adults in Mexico]. Salud Publica Mex. 2013;55 Suppl 2:S323-31. Spanish. PMID 24626711
- [Background] Mazokopakis EE, Starakis IK, Papadomanolaki MG, Mavroeidi NG, Ganotakis ES. The hypolipidaemic effects of Spirulina (Arthrospira platensis) supplementation in a Cretan population: a prospective study. J Sci Food Agric. 2014 Feb;94(3):432-7. doi: 10.1002/jsfa.6261. Epub 2013 Jul 10. PMID 23754631
- [Background] Miczke A, Szulinska M, Hansdorfer-Korzon R, Kregielska-Narozna M, Suliburska J, Walkowiak J, Bogdanski P. Effects of spirulina consumption on body weight, blood pressure, and endothelial function in overweight hypertensive Caucasians: a double-blind, placebo-controlled, randomized trial. Eur Rev Med Pharmacol Sci. 2016;20(1):150-6. PMID 26813468
- [Background] Nagaoka S, Shimizu K, Kaneko H, Shibayama F, Morikawa K, Kanamaru Y, Otsuka A, Hirahashi T, Kato T. A novel protein C-phycocyanin plays a crucial role in the hypocholesterolemic action of Spirulina platensis concentrate in rats. J Nutr. 2005 Oct;135(10):2425-30. doi: 10.1093/jn/135.10.2425. PMID 16177207
- [Background] Petretto DR, Pili R, Gaviano L, Matos Lopez C, Zuddas C. [Active ageing and success: A brief history of conceptual models]. Rev Esp Geriatr Gerontol. 2016 Jul-Aug;51(4):229-41. doi: 10.1016/j.regg.2015.10.003. Epub 2016 May 2. Spanish. PMID 27156859
- [Background] Seo YJ, Kim KJ, Choi J, Koh EJ, Lee BY. Spirulina maxima Extract Reduces Obesity through Suppression of Adipogenesis and Activation of Browning in 3T3-L1 Cells and High-Fat Diet-Induced Obese Mice. Nutrients. 2018 Jun 1;10(6):712. doi: 10.3390/nu10060712. PMID 29865208
- [Background] Serban MC, Sahebkar A, Dragan S, Stoichescu-Hogea G, Ursoniu S, Andrica F, Banach M. A systematic review and meta-analysis of the impact of Spirulina supplementation on plasma lipid concentrations. Clin Nutr. 2016 Aug;35(4):842-51. doi: 10.1016/j.clnu.2015.09.007. Epub 2015 Sep 25. PMID 26433766
- [Background] Szulinska M, Gibas-Dorna M, Miller-Kasprzak E, Suliburska J, Miczke A, Walczak-Galezewska M, Stelmach-Mardas M, Walkowiak J, Bogdanski P. Spirulina maxima improves insulin sensitivity, lipid profile, and total antioxidant status in obese patients with well-treated hypertension: a randomized double-blind placebo-controlled study. Eur Rev Med Pharmacol Sci. 2017 May;21(10):2473-2481. PMID 28617537
- [Background] Torres-Duran PV, Ferreira-Hermosillo A, Juarez-Oropeza MA. Antihyperlipemic and antihypertensive effects of Spirulina maxima in an open sample of Mexican population: a preliminary report. Lipids Health Dis. 2007 Nov 26;6:33. doi: 10.1186/1476-511X-6-33. PMID 18039384
- [Background] Ugwuja E, Ogbonna N, Nwibo A, Onimawo Ia. Overweight and Obesity, Lipid Profile and Atherogenic Indices among Civil Servants in Abakaliki, South Eastern Nigeria. Ann Med Health Sci Res. 2013 Jan;3(1):13-8. doi: 10.4103/2141-9248.109462. PMID 23634323
- [Background] Upasani CD, Balaraman R. Protective effect of Spirulina on lead induced deleterious changes in the lipid peroxidation and endogenous antioxidants in rats. Phytother Res. 2003 Apr;17(4):330-4. doi: 10.1002/ptr.1135. PMID 12722134
- [Derived] Hernandez-Lepe MA, Manriquez-Torres JJ, Ramos-Lopez O, Serrano-Medina A, Ortiz-Ortiz M, Aburto-Corona JA, Pozos-Parra MDP, Villalobos-Gallegos LE, Rodriguez-Uribe G, Gomez-Miranda LM. Impact of Spirulina maxima Intake and Exercise (SIE) on Metabolic and Fitness Parameters in Sedentary Older Adults with Excessive Body Mass: Study Protocol of a Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Feb 8;18(4):1605. doi: 10.3390/ijerph18041605. PMID 33567780